CLINICAL TRIAL: NCT02158754
Title: Clinician Utilization of Corus CAD (or ASGES) in Primary Care Provider Decision Making
Acronym: CU-PCP
Status: Withdrawn | Type: Observational
Why Stopped: Study halted due to low investigator involvement; no patients enrolled in study.
Sponsor: CardioDx (Industry)
Responsible Party: Sponsor
Other Study IDs: CDX_000021; CU-PCP (Other: CardioDx)
Record Dates: First submitted 2014-06-05; First posted 2014-06-09 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease; Angina Pectoris; Chest Pain; Cardiovascular Diseases; CAD; CVD; Coronary Heart Disease; CHD
Keywords: Corus CAD; ASGES; Coronary Artery Disease; Gene Expression; Age/Sex/Gene Expression Score; GES; Angina Pectoris; Chest Pain; Cardiovascular Disease; CAD; CVD; CHD; Coronary Heart Disease; Precision Medicine; Clinical Utility
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Chest Pain; Cardiovascular Diseases; Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Corus CAD (ASGES): Subjects receiving CorusCAD (ASGES) gene expression test as part of their diagnostic workup for typical and/or atypical symptoms of obstructive coronary artery disease.
  Interventions: Diagnostic Test: Corus CAD (ASGES)
- Control: Matched subjects in the same practice that did NOT receive Corus CAD (ASGES) as part of their diagnostic workup.

INTERVENTIONS:
Diagnostic Test: Corus CAD (ASGES)
  Groups: Corus CAD (ASGES)

SUMMARY:
This retrospective study will investigate clinician behavior in diagnosing patients with possible obstructive coronary artery disease who received a Corus CAD (Age/Sex/Gene Expression score - ASGES) result compared to patients who did not have the test performed (matched control patients).

DETAILED DESCRIPTION:
This retrospective study will investigate clinician behavior in diagnosing patients with possible obstructive coronary artery disease who received a Corus CAD (Age/Sex/Gene Expression score - ASGES) result compared to patients who did not have the test performed (matched control patients). The data collected will be from primary care practices and will also assess one to two year health outcomes (MACE, procedure complications). Furthermore, in these real world practice settings, the study will investigate the economic impact of Corus CAD (ASGES) usage at each practice using practice specific data, when available.

ELIGIBILITY:
Inclusion Criteria:

For Corus CAD (Age/Sex/Gene Expression score - ASGES) arm:

* Symptoms suggestive of obstructive CAD, according to the opinion of the site clinician
* Age >= 21 years
* Resulted Corus CAD (ASGES) test used during the evaluation and/or diagnosis of symptoms suggestive of obstructive coronary artery disease (CAD), preferably 1 year prior to data collection date.

For Control arm:

* Symptoms suggestive of obstructive CAD, according to the opinion of the site clinician
* Eligible for Corus CAD (ASGES) (see exclusion criteria)
* Matched to Corus CAD (ASGES) patients by sex, age +/-2.5 years, and presenting symptoms

Exclusion Criteria:

* History of myocardial infarction (MI) or CAD prior to the index evaluation
* Presentation of high risk unstable angina for the index evaluation
* Concurrent systemic infection or inflammatory process
* Concurrent MI or acute coronary syndrome
* Known diabetes mellitus diagnosis or laboratory test results suggestive of a diagnosis of diabetes mellitus (e.g., HbA1C >=6.5)
* Use of steroids, immunosuppressive agents, or chemotherapeutic agents, at time of chest pain presentation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a retrospective chart review, in which only de-identified clinical data will be collected and analyzed. The main criterion for inclusion is the occurrence of chest pain (or anginal equivalent) in a subject without known significant CAD or a history of prior myocardial infarction, and the utilization of Corus CAD (Age/Sex/Gene Expression score - ASGES) for the Corus CAD Arm. Additionally, Corus CAD (ASGES) eligible subjects with similar chest pain (or angina equivalent) who did not undergo Corus CAD (ASGES) testing will be included as a control group.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Reduction in advanced cardiac testing in the low Corus CAD (Age/Sex/Gene Expression score - ASGES) score (<=15) group. | 120 days
  The primary endpoint of the study is the change in number of advanced cardiac diagnostic tests (exercise ECG, stress myocardial perfusion imaging (MPI), cardiac computed tomography angiography (CCTA) or invasive coronary angiography (ICA)) ordered and number of subject referrals to specialty care by the primary clinician, comparing low score Corus CAD (<=15) patients (Corus CAD arm) and matched control patients who did not receive Corus CAD testing (control arm).

SECONDARY OUTCOMES:
Tests/referrals ordered, between low score Corus CAD (ASGES) subjects and control subjects | 120 days
  Tests/referrals ordered, between low score Corus CAD (ASGES) subjects and control subjects, allowing for physician-dependent rates.

OTHER OUTCOMES:
Health outcomes ( MACE, procedure complications) between Corus CAD (ASGES) subjects and control subjects, between low score Corus CAD subjects and matched control subjects, and between low score Corus CAD subjects and non-low score Corus CAD subjects | up to 2 years
  Mace and procedure complications will be collected from Corus CAD (ASGES) draw/presentation through date of chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Monane, MD, FACP, Study Chair — CardioDx
Locations (9):
- United States (9):
  - Internet Medical Group, Rutherford, New Jersey
  - Triangle Primary Care, Wake Forest, North Carolina
  - Comprehensive Physicians Associates, LLC, Youngstown, Ohio
  - Northside Medical Center, Youngstown, Ohio
  - J. Frank Martin, LLC, Columbia, South Carolina
  - South Carolina Internal Medicine Associates LLC, Irmo, South Carolina
  - Colonial Family Practice, Sumter, South Carolina
  - Bells Medical Clinic, Bells, Texas
  - Texas Familicare, Hurst, Texas